CLINICAL TRIAL: NCT05966012
Title: Are Higher Doses of Tranexamic Acid Associated With a Lower Incidence of Post-operative Delirium After Cardiac Surgery? A Retrospective Cohort Study
Brief Title: Tranexamic Acid Dose and Confusion After Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: IRAS 323740
Record Dates: First submitted 2023-07-13; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Cardiovascular Surgery
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Tranexamic acid — Recent data suggests that antifibrinolytics like tranexamic acid (TXA) might be able to lessen the inflammation of the nervous system caused by surgery and CPB through the inhibition of plasmin production, thereby stabilising the blood brain barrier.

SUMMARY:
Delirium is one of the most common complications after cardiac surgery and occurs with an incidence of 3 - 70%.

Both predisposing factors (age, diabetes, severity of cardiac disease, atrial fibrillation) and precipitating factors (type of surgery, duration of cardiopulmonary bypass (CPB) and surgery, ventilator time in ICU, highest temperature in intensive care (ICU)) are difficult to influence. Post-operative delirium is a devastating complication, leading to longer ICU and hospital stay, increased incidence of discharge to nursing facility and poorer long-term cognitive outcome.

Despite the impact this complication has on individuals, their families and healthcare resources, little is known about the causes and potential preventative measures.

It is thought that systemic inflammation compromising the integrity of the blood brain barrier is an important contributing factor. Recent data suggests that antifibrinolytics like tranexamic acid (TXA) might be able to lessen the inflammation of the nervous system caused by surgery and CPB through the inhibition of plasmin production, thereby stabilising the blood brain barrier. Worldwide, the use of TXA has become standard of care in cardiac surgery and other types of surgery with a high risk of bleeding. It has been shown to reduce bleeding by 25% and significantly reduce the rate of transfusion in cardiac and noncardiac surgery.

At Royal Papworth hospital it is routine practice to administer 2g of TXA before commencing CPB irrespective of patients' body weight. We are hypothesising that there is a weight-based effect of TXA on neurological outcomes after cardiac surgery, showing a signal that a higher dose per kg bodyweight will lead to less delirium measured with the Richmond Agitation-Sedation Score (RASS). We intend to analyse 4 years' worth of patient data (05/2018 - 08/2022); the necessary information is routinely collected on using the hospital anaesthetic and ICU record.

DETAILED DESCRIPTION:
There will be no patient contact at any point of this retrospective analysis. The data collected will have been routinely collected on the hospital's electronic systems as part of routine clinical care and data collection.

This is a very new field of interest in cardiac anaesthesia / surgery. No clinical data is currently available apart from recent preliminary data suggesting that Tranexamic Acid (TXA) improves the inflammatory reaction the nervous system has to surgery and cardiopulmonary bypass. The first trial in this area, a RCT (TXA vs no TXA) in abdominal surgery, has only just started recruiting (Tranexamic Acid to Reduce Delirium After Gastrointestinal Surgery: the TRIGS-D Trial; clinicaltrials.gov).

The statistical methods will be determined once data distribution is known; the interdependence of primary and secondary outcome measures will be determined by multivariate regression analysis.

At this stage it is not possible to devise a prospective randomised controlled trial similar the TRIGS-D study in cardiac surgery as giving TXA is considered standard of care. It might be possible, however, to design a RCT comparing different TXA dosing regimens once the the results of this retrospective analysis are available.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing elective or in-house urgent cardiac surgery at RPH between 05/2018 and 08/2022

Exclusion Criteria:

Patients undergoing

* operations involving deep hypothermic circulatory arrest,
* operations involving thoracic vessels other than the ascending aorta,
* solid organ transplantation or mechanical assist device implantation,
* emergency operations

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing elective or in-house urgent cardiac surgery at RPH between 05/2018 and 08/2022
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Richmond Agitation Sedation Score | Up to 48hours after surgery

SECONDARY OUTCOMES:
30 day mortality | Up to 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No